CLINICAL TRIAL: NCT05895864
Title: Utidelone Treated for the Recurrent or Metastatic Urothelial Carcinoma After Prior Chemotherapy: a Open-label, Multicenter Phase II Study (UTRUST)
Brief Title: Utidelone Treated for the Recurrent or Metastatic Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-515-02
Record Dates: First submitted 2023-02-19; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: Drug: Utidelone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Utidelone (Experimental): Utidelone Injection: 35 mg/m2/day, IV on day 1-day 5 of each 21 day cycle, administered to enrolled patients with recurrent or metastatic urothelial carcinoma Number of Cycles: until progression or unacceptable toxicity develops or up to 8 cycles.
  Interventions: Drug: utidelone injection

INTERVENTIONS:
Drug: utidelone injection — utidelone monotherapy in patients with recurrent or metastatic urothelial carcinoma by utidelone
  Other Names: UTD1 injection

SUMMARY:
This study is a open-label, multicenter, phase II study to evaluate the efficacy and safety of utidelone in the recurrent or metastatic urothelial carcinoma after prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years
2. Histologically confirmed urothelial carcinoma (pelvis, ureter, bladder, urethra)
3. Recurrent (unresectable) or metastatic urothelial carcinoma, Patients with primary urothelial carcinoma, mixed with other tissue components, failed or intolerant to standard treatment, and failed to receive neoadjuvant chemotherapy combined with immunotherapy for 12 months were allowed
4. At least one measurable disease according to the response evaluation criteria in solid tumor (RECIST 1.1)
5. Eastern Cooperative Oncology Group (ECOG) performance status between 0 and 2
6. The results of patient's laboratory biochemistry tests are as follows:

   * Normal blood routine within 1 week before enrollment (no blood transfusion or hematopoietic stimulating factor therapy within 14 days) :Hemoglobin(Hb) ≥ 90g/L; Neutrophil count (ANC) > 1.5x109 / L; Platelet count (PLT) ≥ 75×109/L
   * Renal function: serum creatinine ≤ normal upper limit (ULN)
   * Liver and renal function:

   Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT)≤ 3 x ULN, total bilirubin ≤1.5 x ULN, Serum creatinine :≤1.5× ULN or creatinine clearance (Ccr)≥50 ml/min
7. Life expectancy ≥ 3 months
8. Male or female patients of child-producing potential must agree to use double barrier contraception, oral contraceptives, or avoidance of pregnancy measures during the study and for 3 months after the last day of treatment.
9. Females of childbearing potential must have a negative serum pregnancy test at screening and must agree to use double barrier contraception, oral contraceptives, or avoidance of pregnancy measures during the study and for 6 months after the last day of treatment.

Exclusion Criteria:

1. Pregnant or lactating women
2. Suitable for radical means with a chance of cure
3. Patients had received radiation therapy, TKI, or immune checkpoint inhibitor within 2 weeks after the initiation of the study
4. Major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to initial use of the study drug
5. Received an investigational agent, chemotherapy, biological therapy, hormonal therapy, targeted therapy, or radiotherapy within 30 days prior to commencing study treatment, or have not recovered from all treatment-related toxicities to Common Toxicity Criteria (CTC) Grade less than or equal to 1, except for alopecia.CTCAE v.5.0 Grade greater than or equal to 2 peripheral neuropathy;
6. Known active infection with human immunodeficiency virus (HIV), hepatitis B, virus (HBV) or hepatitis C; virus (HCV)
7. Prior allergies to castor oil
8. Patients with symptomatic central nervous system metastases are not permitted, except for those with stable and asymptomatic brain metastases who have completed cranial irradiation, and have at least one measurable lesion outside the brain. Radiotherapy should be completed within 4 weeks prior to the registration
9. Patients with mental disorders or poor compliance
10. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, degree II-III atrioventricular block, etc. The mean QTcF obtained from three 12-lead ECG examinations at rest was >470ms. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular events occurred within 6 months before the first dose of dose. Clinically uncontrolled hypertension
11. Subjects with any other conditions were considered unfit for this study determined by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-06-07 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-13 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 24 months
  Reflected by percentage of tumor size reduction or regression, assessed by imaging techniques and expressed as Objective Response Rate (ORR）

SECONDARY OUTCOMES:
Clinical Benefit Rate | 24 weeks
  CR,PR and SD greater than or equal to 24 weeks
Progression Free Survival (PFS) | 24 months
  Time from date of administration of Utidelone to progression or death
Adverse Events and Serious Adverse Events Safety | up to 3 years
  The incidence of grade ≥3 adverse reactions and the improvement of quality of life were observed

CONTACTS AND LOCATIONS:
Overall Officials: Herui Yao, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Tianxin Lin, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China